CLINICAL TRIAL: NCT03069495
Title: Role of Circulating Innate Lymphoid Cells in Allergic Disorders
Status: Terminated | Type: Observational
Why Stopped: Lack of research assistant to work on study
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0197-17-EP
Record Dates: First submitted 2017-02-22; First posted 2017-03-03 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Allergy; Asthma; Urticaria
Keywords: Allergy; Asthma; Urticaria
MeSH Terms: conditions — Hypersensitivity; Asthma; Urticaria

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — A one time blood draw
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Control Adult Subjects: Healthy adult subjects between the ages of 19-50 years will be enrolled.
- Asthmatic Adult Subjects: Adult subjects between the ages of 19-50 years with mild-to-moderate asthma seen within the UNMC Allergy and Pulmonary Clinics will be invited to be enrolled.
- Chronic Urticaria Adult Subjects: Adult subjects between the ages of 19-50 years with chronic urticaria seen within the UNMC Allergy Clinics will be invited to be enrolled.

SUMMARY:
This study evaluates blood type 2 innate lymphoid cells in participants with mild to moderate asthma and participants with chronic urticaria as compared to healthy adult participants.

DETAILED DESCRIPTION:
The first objective of this study is to determine whether blood ILC2s differ in female vs. male allergic asthmatics. This is because females become more susceptible to asthma after puberty and experience more severe disease as adults.

The second objective of this study is to determine whether ILC2 cells in chronic urticaria differ from healthy controls.

There will be one shared healthy control adult subject group for comparison for objective 1 and 2.

In this study, there will be a blood draw once on 3 different adult populations aged 19-50 years: 1) Participants with mild-to moderate allergic asthma; 2) Participants with chronic urticaria, and 3) Healthy control adult participants. Demographics and allergy indicators will be collected from the medical chart. The investigators will acquire whole blood for serum and acquisition of specific lymphocyte populations. There will be no intervention or research follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects between age 19-50 years.
2. Non-smokers, defined as < 100 cigarettes in lifetime.

Exclusion Criteria:

1. Female donors will be excluded if they are menopausal or have undergone total abdominal hysterectomy and/or bilateral salpingoophorectomy
2. For female donors, blood draw cannot occur during menstrual period time. Subjects will be excluded if they have menstrual period at timing of blood draw.
3. Current and past smokers.
4. Subjects with asthma and any other lung disease including chronic obstructive pulmonary disease, interstitial lung disease, pulmonary hypertension, sarcoidosis, cystic fibrosis.
5. Pregnant or lactating subjects
6. Subjects with hypercalcemia (> 10.3 mg/dL), renal insufficiency (glomerular filtration rate [GFR] < 50 mL/min/1.73m2), or malignancy.
7. Subjects with any symptoms of respiratory infection in the past 4 weeks.
8. Subjects unable to hold leukotriene modifiers or antihistamines for at least 24 hours prior to blood draw.
9. Subjects on any immunomodulators, including omalizumab, or systemic corticosteroid in the past 4 weeks.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult subjects age 19-50 years.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
ILC2 Phenotype | 52 weeks
  Blood ILC2s responsiveness will be determined solely for research purposes using ex vivo stimulation assays.

CONTACTS AND LOCATIONS:
Overall Officials: Jill A Poole, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
Subject information will be de-identified. IPD will not be made available to other researchers.